CLINICAL TRIAL: NCT02362854
Title: A Randomized Clinical Trial of an Adjunct Diode Laser Application in the Treatment of Peri-implantitis.
Brief Title: Efficacy of Diode Laser in Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University Research Fund (Unknown)
Responsible Party: Principal Investigator, Volkan Arisan, Assoc.Prof.Dr, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulU
Record Dates: First submitted 2014-09-16; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Implant; Peri-Implantitis; Alveolar Bone Loss; Complications
Keywords: dental implant; laser; diode laser; peri-implantitis; bacterial count
MeSH Terms: conditions — Peri-Implantitis; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional peri-implantitis treatment (Active Comparator): Peri-implantitis treatment according to the Cumulative interceptive supportive (CIST) therapy.
  Interventions: Procedure: Conventional peri-implantitis treatment
- DL application in peri-implantitis (Experimental): Adjunct Diode Laser application.
  Interventions: Device: DL application in peri-implantitis

INTERVENTIONS:
Procedure: Conventional peri-implantitis treatment — Elimination of the bacterial plaque. Establishing optimal healing conditions. Detoxification of the affected environment.
  Other Names: CIST treatment protocol
  Arms: Conventional peri-implantitis treatment
Device: DL application in peri-implantitis — Diode laser application in the diseased implants.
  Arms: DL application in peri-implantitis

SUMMARY:
The aim of this study was to compare the efficacy of a diode laser (DL) as an adjunct to conventional scaling in the treatment of mild-to-moderate peri-implantitis. A prospective clinical, radiographic and microbiologic split-mouth study was conducted to test the following null hypothesis; adjunct application of a diode laser, in the conventional treatment of peri-implantitis, are not associated with a statistically significant difference regarding the microbial counts, marginal bone loss and peri-implant parameters.

DETAILED DESCRIPTION:
Efficacy of a diode laser (DL) in peri-implantitis was investigated. 48 implants diagnosed with peri-implantitis were included. In addition to the conventional scaling and debridement, random 24 implants were lased by a DL. Periodontal indexes, microbiologic specimens and radiographs were used for assessment. Baseline parameters were similar between groups. After six months laser group revealed higher MBL than the control group. Microbiota of the implants were found unchanged after one month. DL appears to have no additional positive influence on the peri-implantitis treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* No local and systemic health problems prohibit the study interventions
* Bi-lateral implants with peri-implantitis diagnosis

Exclusion Criteria:

* Local and systemic health problems prohibiting the study interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bacterial counts | One month
  Bacterial load around the the diseased implants will be determined at the initiation of the study. The assessment will be performed after one months

SECONDARY OUTCOMES:
Marginal Bone loss | Six months
  The marginal bone loss around the diseased implants will be assessed after six months to analyse any bone level change.

OTHER OUTCOMES:
Peri-implant health indexes | one and six months
  Bleeding on probing, probing depth and plaque index which determined at the initiation of the study will be re-evaluated after one and six months to asees the effect of the variables

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Arısan, Ass.Prof.Dr., Study Chair — Istanbul University, Faculty of Dentistry; Cuneyt Karabuda, Prof.Dr., Study Director — Istanbul University, Faculty of Dentistry
Locations (1):
- Department of Oral Implantology, Faculty of Dentistry, Istanbul University, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- See also: Department web link — http://dishekimligi.istanbul.edu.tr/oral-implantoji/